CLINICAL TRIAL: NCT02756364
Title: An Open-Label Phase 2 Study of MLN0128 (A TORC1/2 Inhibitor) in Combination With Fulvestrant in Women With ER-Positive/HER2-Negative Advanced or Metastatic Breast Cancer That Has Progressed During or After Aromatase Inhibitor Therapy
Brief Title: Sapanisertib in Combination With Fulvestrant in Women With Advanced or Metastatic Breast Cancer After Aromatase Inhibitor Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C31006; 2015-003612-20 (EudraCT Number); U1111-1174-2165 (Registry Identifier: WHO)
Record Dates: First submitted 2016-04-28; First posted 2016-04-29 (Estimated); Results first posted 2020-12-19 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Breast Neoplasms
Keywords: Drug Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fulvestrant 500 mg (Active Comparator): Fulvestrant 500 mg, intramuscularly (IM), once on Days 1 and 15 in Cycle 1, and then on Day 1 of each subsequent 28-day cycle until progressive disease, unacceptable toxicity, or withdrawal of consent (Median duration of treatment was 16.0 weeks).
  Interventions: Drug: Fulvestrant
- Fulvestrant 500 mg + Sapanisertib 4 mg (Experimental): Fulvestrant 500 mg, IM, once on Days 1 and 15 in Cycle 1, and then on Day 1 of each subsequent 28-day cycle along with the sapanisertib 4 mg, capsules, orally, once daily in each 28-day treatment cycle until progressive disease, unacceptable toxicity, or withdrawal of consent (Median duration of treatment was 20.1 and 20.3 weeks for fulvestrant and sapanisertib respectively).
  Interventions: Drug: Fulvestrant; Drug: Sapanisertib
- Fulvestrant 500 mg + Sapanisertib 30 mg (Experimental): Fulvestrant 500 mg, IM, once on Days 1 and 15 in Cycle 1, and then on Day 1 of each subsequent 28-day cycle along with sapanisertib 30 mg, capsule, orally, once weekly in each 28-day treatment cycle until progressive disease, unacceptable toxicity, or withdrawal of consent (Median duration of treatment was 17.0 weeks for fulvestrant and sapanisertib, each).
  Interventions: Drug: Fulvestrant; Drug: Sapanisertib

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant IM injection.
Drug: Sapanisertib — Sapanisertib capsule.
  Other Names: MLN0128
  Arms: Fulvestrant 500 mg + Sapanisertib 30 mg; Fulvestrant 500 mg + Sapanisertib 4 mg

SUMMARY:
The primary purpose of this study is to compare the progression free survival (PFS) of participants treated with the combination of fulvestrant plus daily sapanisertib and fulvestrant plus weekly sapanisertib versus participants treated with single-agent fulvestrant.

DETAILED DESCRIPTION:
The drug being tested in this study is called sapanisertib. Sapanisertib is being tested to treat postmenopausal women with advanced or metastatic estrogen receptor (ER) positive, human epidermal growth factor receptor-2 (HER2) negative breast cancer that has progressed during or after aromatase inhibitor (AI) therapy. This study will evaluate the efficacy and safety of combination of fulvestrant + daily sapanisertib and fulvestrant + weekly sapanisertib compared with fulvestrant alone.

The study will enroll approximately 153 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the three treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Fulvestrant 500 mg
* Fulvestrant 500 mg + Sapanisertib 4 mg
* Fulvestrant 500 mg + Sapanisertib 30 mg

All participants will receive either fulvestrant 500 mg intramuscularly (IM), fulvestrant 500 mg + sapanisertib 4 mg daily or fulvestrant 500 mg + sapanisertib 30 mg weekly.

This multicenter trial will be conducted Spain and the USA. Participants will make multiple visits to the clinic, and end of treatment (EOT) visit which will occur 30 to 40 days after receiving their last dose of study drug or before the start of any subsequent anticancer therapy. After EOT, participants will be followed for progression free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Female participants aged 18 years or older who are postmenopausal.
2. Histologically proven diagnosis of breast cancer with evidence of metastatic disease or locoregional recurrence.
3. Histological confirmation and documentation of estrogen receptor (ER)-positive status (≥1% positive stained cells).
4. Histological or cytological confirmation and documentation of human epidermal growth factor receptor-2 (HER2)-negative status by local laboratory testing using criteria in the American Society of Oncology (ASCO)/College of American Pathologists (CAP) Clinical Practice Guideline update.
5. Measurable disease defined as either of the following:

   * At least 1 extra-osseous lesion that could be accurately measured in at least 1 dimension.
   * The lesion must have measured ≥20 mm with conventional imaging techniques or ≥10 mm with spiral CT or MRI. Lymph nodes must be ≥1.5 cm in the short axis to be considered measurable.
   * Bone lesions (lytic or mixed [lytic plus sclerotic]) in the absence of measurable disease as defined above. Note: Participants with sclerotic/osteoblastic bone lesions only, in the absence of measurable disease, were not eligible.
6. Progressive Disease (PD) during prior aromatase inhibitor (AI) therapy.
7. Have a history of brain metastasis provided that all of the following criteria are met:

   * Brain metastases have been treated.
   * No evidence of PD for ≥3 months before the first dose of study drug.
   * No hemorrhage after treatment.
   * Off dexamethasone treatment for ≥4 weeks before the first dose of study drug.
   * No ongoing requirement for dexamethasone or anti-epileptic drugs.
8. Eastern cooperative oncology group (ECOG) performance status of 0 or 1.
9. Clinical laboratory values as specified below within 4 weeks before the first dose of study drug:

   * Bone marrow reserve consistent with absolute neutrophil count (ANC) ≥1.5*10^9/L; platelet count ≥100*10^9/L; hemoglobin (Hgb) ≥9 g/dL.
   * Total bilirubin ≤1.5*the upper limit of the normal range (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5*ULN (≤5*ULN if liver metastases are present).
   * Creatinine clearance ≥40 mL/min based on Cockcroft-Gault estimate or based on a 12- or 24-hour urine collection.
   * Fasting serum glucose ≤130 mg/dL and fasting triglycerides ≤300 mg/dL.

Exclusion Criteria:

1. Prior therapy with mechanistic target of rapamycin (mTOR), phosphoinositide-3-kinase (PI3K), or dual PI3K-mTOR inhibitors, serine/threonine-specific protein kinase (AKT) inhibitors, or fulvestrant.
2. Prior treatment with >1 line of chemotherapy for metastatic breast cancer or for locoregional recurrence that was not amenable to resection or radiation therapy with curative intent.
3. Experienced PD on >2 endocrine therapies for metastatic breast cancer or for locoregional recurrence that was not amenable to resection or radiation therapy with curative intent.
4. Life-threatening metastatic visceral disease (defined as extensive hepatic involvement or symptomatic pulmonary lymphangitic spread).
5. Poorly controlled diabetes mellitus defined as hemoglobin A1c (glycosylated hemoglobin; HbA1c) >7%; participants with a history of transient glucose intolerance due to corticosteroid administration may be eligible if all other inclusion/exclusion criteria are met.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal females.
Enrollment: 141 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (53):
- United States (30):
  - Southern Cancer Center, PC, Mobile, Alabama
  - CBCC Global Research 6501 Truxtun Avenue Bakersfield, CA, Bakersfield, California
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - UCSD Moores Cancer Center, La Jolla, California
  - UCLA Hematology/Oncology David Geffen School of Medicine, Los Angeles, California
  - North County Oncology, Oceanside, California
  - Torrance Health Association, Redondo Beach, California
  - PHC-SLO Oncology and Hematology, San Luis Obispo, California
  - Cancer Center of Santa Barbara With Sansum Clinic, Santa Barbara, California
  - University of Colorado Cancer Center-Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - St. Mary'S Hospital Regional Cancer Center, Grand Junction, Colorado
  - Rocky mountain cancer centers LLP, Lakewood, Colorado
  - Holy Cross Hospital- Bienes Cancer Center, Fort Lauderdale, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Orlando Health Inc., Orlando, Florida
  - Ft. Wayne Medical Oncology and Hematology, Inc, Fort Wayne, Indiana
  - New England Cancer Specialists, Scarborough, Maine
  - Health Partners Institute Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - New Jersey Hematology & Oncology Associates, Brick, New Jersey
  - Northern Westchester Hospital Cancer Treatment & Wellness Center, Mount Kisco, New York
  - Oregon Health and Science University, Portland, Oregon
  - Texas Oncology, P.A., Austin, Texas
  - Texas Oncology - Presbyterian Hospital, Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Texas Oncology- South Second Street, McAllen, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology,PA. Tyler TX, 75702, Tyler, Texas
  - Virginia Cancer Specialist PC, Leesburg, Virginia
  - West Virginia University School of Medicine, Morgantown, West Virginia
- Spain (23):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Onkologikoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital Universitario Puerta del Hierro, Majadahonda, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Sant Joan de Reus, Reus, Tarragona
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Centro Oncologico de Galicia, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital De la Santa Creu i Sant Pau, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital General Universitario Morales Messeguer, Murcia
  - Hospital Clinico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen de la Macarena, Seville
  - Fundacion Instituto Valenciano de Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 50 investigative sites in Spain and the United States from 28 July 2016 to 25 November 2019. After all data was collected and participants were transitioned to post-trial access, the Sponsor stopped the study site, defined as 'Site terminated by the Sponsor'.
Pre-assignment Details: Female participants with a diagnosis of estrogen receptor (ER)-positive/human epidermal growth factor receptor-2 (HER2)-negative advanced or metastatic breast cancer that has progressed during or after aromatase inhibitor therapy were enrolled in 1:1:1 ratio to receive fulvestrant, fulvestrant + sapanisertib QD and fulvestrant + sapanisertib QW.
Groups:
- Arm A: Fulvestrant 500 mg: Fulvestrant 500 mg, intramuscularly (IM), once on Days 1 and 15 in Cycle 1, and then on Day 1 of each subsequent 28-day cycle until progressive disease, unacceptable toxicity, or withdrawal of consent (Median duration of treatment was 16.0 weeks).
- Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD: Fulvestrant 500 mg, IM, once on Days 1 and 15 in Cycle 1, and then on Day 1 of each subsequent 28-day cycle along with the sapanisertib 4 mg, capsules, orally, once daily in each 28-day treatment cycle until progressive disease, unacceptable toxicity, or withdrawal of consent (Median duration of treatment was 20.1 and 20.3 weeks for fulvestrant and sapanisertib respectively).
- Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW: Fulvestrant 500 mg, IM, once on Days 1 and 15 in Cycle 1, and then on Day 1 of each subsequent 28-day cycle along with sapanisertib 30 mg, capsule, orally, once weekly in each 28-day treatment cycle until progressive disease, unacceptable toxicity, or withdrawal of consent (Median duration of treatment was 17.0 weeks for fulvestrant and sapanisertib, each).
Period: Overall Study
Arm/Group | Arm A: Fulvestrant 500 mg | Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD | Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW
Started (Full Analysis Set (FAS) - Randomized Participants) | 46 | 47 | 48
Treated Participants (Safety Analysis Set) | 46 | 47 | 47
Completed | 0 | 0 | 0
Not Completed | 46 | 47 | 48
Not completed — Site Terminated by Sponsor | 24 | 30 | 21
Not completed — Death | 20 | 15 | 18
Not completed — Withdrawal by Patient | 2 | 1 | 8
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Fulvestrant 500 mg | Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD | Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW | Total
Number analyzed (Participants) | 46 | 47 | 48 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.10) | 60.3 (10.92) | 57.9 (12.04) | 59.5 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 48 | 141
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 7 | 16
  Not Hispanic or Latino | 37 | 41 | 40 | 118
  Unknown or Not Reported | 4 | 2 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 44 | 45 | 44 | 133
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 23 | 34 | 33 | 90
  United States | 23 | 13 | 15 | 51

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of first documentation of progressive disease (PD) or death due to any cause, whichever occurred first. Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, PD was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Up to 40 months
Population: Full Analysis Set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Fulvestrant 500 mg | Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD | Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW
Number analyzed (Participants) | 46 | 47 | 48
months | 3.5 [1.9 to 5.6] | 7.2 [3.9 to 10.6] | 5.6 [4.1 to 9.0]
Statistical Analysis 1: Comparison: Arm A: Fulvestrant 500 mg vs Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD; Test type: Superiority; p = 0.537, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.47 to 1.26] — HR obtained by stratified Cox proportional hazard model with treatment arm, original interactive response technology (IRT) stratification factors as covariates. A hazard ratio of <1 was considered statistically significant
Statistical Analysis 2: Comparison: Arm A: Fulvestrant 500 mg vs Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW; Test type: Superiority; p = 0.849, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.53 to 1.45] — HR obtained by stratified Cox proportional hazard model with treatment arm, original IRT stratification factors as covariates. A hazard ratio of <1 was considered statistically significant

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death.
Time Frame: Up to 164 weeks
Population: Full Analysis Set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Fulvestrant 500 mg | Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD | Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW
Number analyzed (Participants) | 46 | 47 | 48
months | 30.5 [21.5 to NA] — The upper limit of confidence interval (CI) was not estimable due to fewer number of participants with event. | NA [29.9 to NA] — The median and upper limit of CI was not estimable due to fewer number of participants with event. | 34.2 [20.0 to NA] — The upper limit of CI was not estimable due to fewer number of participants with event.
Statistical Analysis 1: Comparison: Arm A: Fulvestrant 500 mg vs Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD; Test type: Superiority; p = 0.276, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.36 to 1.40] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Arm A: Fulvestrant 500 mg vs Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW; Test type: Superiority; p = 0.470, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.47 to 1.68] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from the date of randomization to the date of first documentation of progression. Per RECIST v1.1, PD was defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Up to 40 months
Population: Full Analysis Set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Fulvestrant 500 mg | Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD | Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW
Number analyzed (Participants) | 46 | 47 | 48
months | 3.5 [1.9 to 5.6] | 7.2 [5.5 to 10.6] | 5.6 [4.1 to 9.0]
Statistical Analysis 1: Comparison: Arm A: Fulvestrant 500 mg vs Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD; Test type: Superiority; p = 0.495, Log Rank; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.46 to 1.25] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Arm A: Fulvestrant 500 mg vs Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW; Test type: Superiority; p = 0.646, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.49 to 1.38] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieve a best response of complete response (CR) or partial response (PR) according to RECIST v1.1 criteria. CR was defined as disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions.
Time Frame: Up to 40 months
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Fulvestrant 500 mg | Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD | Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW
Number analyzed (Participants) | 46 | 47 | 47
percentage of participants | 10.9 | 21.3 | 12.8
Statistical Analysis 1: Comparison: Arm A: Fulvestrant 500 mg vs Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD; Test type: Superiority; Odds Ratio (OR) = 2.23, 95% CI 2-sided [0.68 to 7.29] — The odds ratio and 95% CIs were obtained using a stratified Cochran-Mantel-Haenszel model with the original IRT stratification factors (visceral metastases, previous sensitivity to hormonal therapy, and previous exposure to CDK4/6 inhibitors)
Statistical Analysis 2: Comparison: Arm A: Fulvestrant 500 mg vs Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW; Test type: Superiority; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.34 to 4.39] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants who achieved a best response of CR, PR, or stable disease (SD) of any duration. CR was defined as disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Up to 40 months
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Fulvestrant 500 mg | Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD | Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW
Number analyzed (Participants) | 46 | 47 | 47
percentage of participants | 60.9 | 74.5 | 66.0
Statistical Analysis 1: Comparison: Arm A: Fulvestrant 500 mg vs Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD; Test type: Superiority; Odds Ratio (OR) = 2.56, 95% CI 2-sided [0.94 to 6.94] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Fulvestrant 500 mg vs Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW; Test type: Superiority; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.69 to 4.44] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Percentage of Participants Who Experienced at Least One Treatment-emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Up to 164 weeks
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Fulvestrant 500 mg | Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD | Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW
Number analyzed (Participants) | 46 | 47 | 47
percentage of participants | 89.1 | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: Up to 164 weeks
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. All-cause Mortality or data for deaths were collected in FAS population. Adverse events were collected in Safety Analysis Set.
Arm/Group | Arm A: Fulvestrant 500 mg | Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD | Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW
All-Cause Mortality (participants affected / at risk) | 20/46 | 15/47 | 18/48
Serious Adverse Events (participants affected / at risk) | 8/46 | 13/47 | 8/47
Other Adverse Events (participants affected / at risk) | 38/46 | 47/47 | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Fulvestrant 500 mg (N=46) | Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD (N=47) | Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW (N=47)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 2
Appendicitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Fulvestrant 500 mg (N=46) | Arm B: Fulvestrant 500 mg + Sapanisertib 4 mg QD (N=47) | Arm C: Fulvestrant 500 mg + Sapanisertib 30 mg QW (N=47)
Nausea (Gastrointestinal disorders) | 9 | 23 | 41
Vomiting (Gastrointestinal disorders) | 4 | 14 | 33
Diarrhoea (Gastrointestinal disorders) | 1 | 24 | 13
Stomatitis (Gastrointestinal disorders) | 3 | 16 | 15
Constipation (Gastrointestinal disorders) | 8 | 4 | 6
Dry mouth (Gastrointestinal disorders) | 1 | 12 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5 | 9
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 3
Gastritis (Gastrointestinal disorders) | 0 | 3 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 3
Asthenia (General disorders) | 11 | 13 | 21
Fatigue (General disorders) | 10 | 17 | 11
Pyrexia (General disorders) | 3 | 4 | 4
Injection site pain (General disorders) | 5 | 2 | 2
Malaise (General disorders) | 0 | 1 | 4
Pain (General disorders) | 1 | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 27 | 26
Decreased appetite (Metabolism and nutrition disorders) | 5 | 15 | 19
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 6 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Headache (Nervous system disorders) | 9 | 4 | 10
Dysgeusia (Nervous system disorders) | 0 | 8 | 7
Dizziness (Nervous system disorders) | 1 | 4 | 5
Somnolence (Nervous system disorders) | 0 | 4 | 0
Tremor (Nervous system disorders) | 0 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 15 | 8
Rash (Skin and subcutaneous tissue disorders) | 0 | 14 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Weight decreased (Investigations) | 1 | 11 | 6
Aspartate aminotransferase increased (Investigations) | 2 | 6 | 6
Alanine aminotransferase increased (Investigations) | 2 | 6 | 4
Gamma-glutamyltransferase increased (Investigations) | 1 | 5 | 3
Blood cholesterol increased (Investigations) | 0 | 5 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 3 | 1
Neutrophil count decreased (Investigations) | 0 | 3 | 2
Urinary tract infection (Infections and infestations) | 2 | 7 | 7
Nasopharyngitis (Infections and infestations) | 4 | 5 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 5 | 1
Respiratory tract infection (Infections and infestations) | 3 | 2 | 1
Anxiety (Psychiatric disorders) | 5 | 5 | 2
Depression (Psychiatric disorders) | 3 | 4 | 3
Insomnia (Psychiatric disorders) | 0 | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 1
Hypertension (Vascular disorders) | 7 | 4 | 5
Hot flush (Vascular disorders) | 5 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 2
Dysuria (Renal and urinary disorders) | 0 | 2 | 3
Tinnitus (Ear and labyrinth disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT02756364/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT02756364/SAP_001.pdf